CLINICAL TRIAL: NCT06424561
Title: The Influence of Systematic Psychological Intervention on Patients Undergoing VSD Drainage Surgery for Chronic Infected Wounds
Brief Title: The Influence of Systematic Psychological Intervention on Patients About VSD Drainage Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-2024-085
Record Dates: First submitted 2024-05-03; First posted 2024-05-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Chronic Wounds
Keywords: VSD drainage surgery; systematic psychological intervention; chronic wounds

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Intervention Group (Experimental): The patients in the intervention group received systematic psychological intervention on the basis of routine nursing after admission, the main steps were as follows: 1 preoperative and postoperative psychological assessment (self-rating anxiety scale (SAS) and self-rating depression scale (SDS-RRB- to assess the psychological status of patients) , this part through medical records, face-to-fAssessmentment and questionnaire survey; Timely attention to patients' psychological state. 2 at the end of the evaluation, we can start the psychological intervention, collect the pre-intervention scale and post-intervention scale, collect the data, and make records according to the collected data, so as to carry on the follow-up work in the later period. 3 the days of hospitalization, the satisfaction of hospitalization, the expenses of hospitalization and the psychological scale were recorded, and the influence of psychological intervention on the patients was compared with the routine group.
  Interventions: Behavioral: Psychological Intervention Group
- Routine care group (No Intervention): Routine nursing care is carried out by the regular group based on the measures for VSD drainage procedure.

INTERVENTIONS:
Behavioral: Psychological Intervention Group — The intervention group provides psychological education to patients, emphasizing participation in a "Surgery Success" patient group organized by researchers, and collects successful patient cases for promotion. Patients are encouraged to learn from successful cases within the group. Psychological intervention is also provided to family members, as they are the primary caregivers, and guiding their thoughts is crucial. Timely identification of patients with psychological abnormalities is conducted, with psychological consultations if necessary. Targeted measures are taken for patients with psychological abnormalities. Upon discharge, one-on-one consultation and tracking services are provided by designated nurses to alleviate patients' feelings of helplessness and despair, continuing until the patient fully recovers.
  Other Names: Experimental group
  Arms: Psychological Intervention Group

SUMMARY:
This study focuses on providing clinical care to patients undergoing VSD drainage surgery for chronic wounds, while also paying attention to the impact of negative emotions such as depression and anxiety, as well as quality of life and social support, on the patients' physical and mental well-being. It observes the influence of psychology on patients.

DETAILED DESCRIPTION:
The chronic, difficult-to-heal wounds not recovering within the expected timeframe not only impact the quality of life for patients and hinder the recovery of the primary condition but also exacerbate their financial and psychological burdens, further affecting the quality of wound healing. The objective of this study is to employ psychological nursing interventions effectively combined with nursing techniques and communication strategies. By listening to patients' fears, anxieties, and tensions, it significantly alleviates their negative emotions, enhances compliance with medical advice, and predicts postoperative complications to mitigate them. Tailored and empathetic care, along with psychological counseling, is provided to expedite wound healing.

ELIGIBILITY:
Inclusion Criteria:

- A mentally healthy, communicative adult. Patients and their families are cooperative, understanding, and supportive of this study.

Adult patients undergoing VSD surgery for chronic wounds.

Exclusion Criteria:

- Patients who are unable to effectively cooperate with nursing questionnaires due to auditory or visual impairments, cognitive impairments, or low levels of cultural literacy.

Patients with poor compliance or those who harbor skepticism and hostility towards this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-rating anxiety scale (SAS) | After 4 weeks of intervention
  The Self-Rating Anxiety Scale (SAS) was developed by W.K. Zung in 1971. This scale consists of 20 items reflecting subjective feelings of anxiety, with each item rated on a four-point scale based on the frequency of symptoms. The scoring criteria are as follows: "1" indicates none or very little time; "2" indicates some of the time; "3" indicates a good part of the time; "4" indicates most or all of the time.According to normative results, in China, the standard deviation cutoff for SAS is 53 points. The divisions are as follows:53 to 62 points: Mild anxiety，63 to 72 points: Moderate anxiety，Above 72 points: Severe anxiety.
self-rating depression scale (SDS） | After 4 weeks of intervention
  The Self-Rating Depression Scale (SDS) was developed by W.K. Zung in 1965. This scale comprises 20 items reflecting subjective feelings of depression, with each item rated on a four-point scale based on the frequency of symptoms. For positively scored items, the ratings are 1, 2, 3, 4 respectively, while for negatively scored items, they are 4, 3, 2, 1. The normal upper limit for the total raw score of SDS is 41 points, with lower scores indicating better states. The standard score is obtained by multiplying the total raw score by 1.25 and taking the integer part. The standard deviation cutoff for SDS is 53 points. The divisions are as follows:53 to 62points:Mild depression，63 to 72 points: Moderate depression，Above 73 points: Severe depression.

SECONDARY OUTCOMES:
Patient satisfaction with hospitalization | After 4 weeks of intervention
  The satisfaction was calculated using our hospital's unified discharge satisfaction questionnaire for inpatients. Each item is rated on a scale of 1 to 5, with a total of 20 items and a maximum score of 100 points. Scores above 95 are considered satisfied, scores between 90 and 95 are deemed basically satisfied, and scores below 90 indicate dissatisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No